## **Note on Registration Timing:**

This study was initiated on 30-1-2024. Initially, I was not aware of the importance of early registration on ClinicalTrials.gov. Registration was completed after the study began to ensure transparency and adherence to ethical guidelines. All study procedures and protocols have been conducted under the supervision of the academic advisor.

Republic of Yemen
Sana'a University
Faculty of Dentistry
Postgraduate Studies and Scientific Research
Department of Orthodontics Pedodontics and Preventive Dentistry
Orthodontics Program



## **Consent Form**

I'm .....agree to participate in this research named

| Evaluation of the Effectiveness of Elastic chains Versus Elastics on Maxillary Canine<br>Retraction: A Randomized Clinical Trial |
|---|
| I know that I will be one of the volunteers who will be studied. I also know that x-rays and study models will be taken prior and after teeth retraction. |
| Being a volunteer or refusal to participate in this study will have no effected from any person. |
| The risk associated with being volunteer is absent. Data and information I give will be confidential and used only for medical research purpose. |
| I understand that my name will not be used as in any scientific publication and that my privacy will be strictly maintained. I may withdraw from this study at any time. |
| Date: |
| Signature of participant: |